CLINICAL TRIAL: NCT03792867
Title: Radical Resection and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in the Treatment of High Risk Recurrent Retroperitoneal Sarcoma
Brief Title: Radical Resection and HIPEC for Recurrent Retroperitoneal Sarcoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/2012/B
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Retroperitoneal Sarcoma
MeSH Terms: interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radical Resection and HIPEC (Experimental)
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — Immediately after resection, 15mg/m2 doxorubicin will be administered by peritoneal perfusion for 60 minutes and then drained.

SUMMARY:
Retroperitoneal sarcoma is a rare cancer that accounts for 15% of soft tissue sarcomas and affects many young people. In approximately 50% of patients, the tumour will reappear in the same area regardless of therapy. Current treatment involves radical resection; however, it does not significantly reduce recurrence rates or improve overall survival. Recurrent retroperitoneal sarcoma does not respond well to chemotherapy and prognosis is often guarded. One of the main challenges in the surgical treatment of this disease is the ability to accurately identify the local extension of the disease and to prevent local recurrence.

At present, there are no options to prevent recurrence after surgery. In recent years, there has been increased interest in the use of combined radical surgery with heated intraperitoneal chemotherapy (HIPEC). Radical resection is defined as en-bloc resection of the tumour including but not limited to surrounding organ resection and normal fat. This is in combination with the use of HIPEC. HIPEC is the use of chemotherapy in the intraperitoneal cavity that is heated to 40 to 42 degree Celsius.

Surgery coupled with HIPEC has shown to reduce recurrence in colorectal cancer, appendiceal cancer and mesothelioma. We hypothesize that HIPEC when coupled with radical surgery will improve the overall outcomes of patients with retroperitoneal sarcomatosis. We hope to learn if this treatment approach will increase locoregional control to reduce recurrence rates and improve survival.

ELIGIBILITY:
Inclusion Criteria:

1. Disease Characteristics

   1. Histologically proven soft tissue sarcoma of one of following high-risk groups:

      * Tumours with grade 2 or 3 histology
      * Size more than or equal to 5cm
      * Extracompartmental and deep extension
   2. Local recurrence of primary tumour
   3. Inadequate surgical excision of previously operated on tumour
   4. Proven diagnosis of recurrent retroperitoneal sarcoma confirmed by imaging modality and/ or intraoperative biopsy
2. Patient Characteristics

   1. Age: ≥21 years old
   2. Performance status: ECOG 0-1
   3. Normal haematological, hepatic, coagulation, renal and electrolyte profiles
   4. Normal left ventricular ejection fraction
   5. Not pregnant or nursing

Exclusion Criteria:

1. Patient is medically unfit for surgery due to concurrent medical comorbidities.
2. Any medical or psychiatric condition(s) which would preclude informed consent.
3. Patient is pregnant or nursing.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | From time of resection to one year post-surgery
  To evaluate chemotherapy toxicity and unforeseen acute and late complications associated with the treatment

SECONDARY OUTCOMES:
Local recurrence-free survival | From time of resection until first occurrence of disease recurrence, up to 3 years
  To determine if the introduction of radical surgery and HIPEC would improve the local recurrence-free survival of patients as compared to current treatment strategies
Overall survival | From time of resection to death from any cause, up to 3 years
  To determine if the introduction of radical surgery and HIPEC would improve the overall survival of patients as compared to current treatment strategies

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Ong, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seo CJ, Tan JW, Farid M, Wong JSM, Soo KC, Chia CS, Ong CJ. Radical resection and hyperthermic intraperitoneal chemotherapy (HIPEC) in the treatment of high risk recurrent retroperitoneal sarcoma-A pilot study in a tertiary Asian centre. PLoS One. 2024 Apr 4;19(4):e0300594. doi: 10.1371/journal.pone.0300594. eCollection 2024. PMID 38574044